CLINICAL TRIAL: NCT01302002
Title: The Use of Metformin in Early Breast Cancer Patients Pre-Surgery: A Phase 0 Study Regarding The Biological Effect
Brief Title: The Use of Metformin in Early Breast Cancer Patients Pre-Surgery
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Ana Elisa Lohmann, Medical Oncologist, Instituto Nacional de Cancer, Brazil
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INCA113/10
Record Dates: First submitted 2011-02-14; First posted 2011-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metformin; Pre-Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin Pre-Surgery (Experimental): Patients will take metformin twice a day for three weeks prior surgery
  Interventions: Drug: Metformin Pre-Surgery

INTERVENTIONS:
Drug: Metformin Pre-Surgery — 500 mg tablet, taken twice a day for 3 weeks
  Other Names: Laboratory biomarker analysis; Blood and tissue collection

SUMMARY:
The study will test metformin in patients with early breast cancer. Blood and tissue will be collected before and after the use of metformin.

DETAILED DESCRIPTION:
Patients will take metformin twice a day for 3 weeks before surgery. The hypothesis is that metformin will reduce cell proliferation rates (Ki67) and increase apoptoses (TUNEL)in tumor tissue.

The study will collect and analyze pre- and post-treatment blood specimens for:

* Serum glucose
* Insulin levels
* Estradiol
* HOMA test
* Glycosylated haemoglobin

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer T1 or T2, Nx
* Knowledge of the investigational nature of the study and ability to provide consent for study participation

Exclusion Criteria:

* Diabetes or baseline glucose or Glycosylated haemoglobin upper limit of normal for the institution
* Recent use of corticosteroids
* AST > 1.5 times upper limit of normal for the institution
* Pregnancy
* Serious clinical illness
* Prior or concurrent systemic neoadjuvant Breast Cancer therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To determine the in situ effects of metformin in women with operable stage I or II breast cancer | 60 days after the surgery
  To determine the in situ effects of metformin on
  * proliferation (Ki67) and apoptosis (TUNEL), fosforilate AKT
  * CD1a CD83, CD68, F40/80, arginase iNOS and T cells -CD4(+),CD45RA(+), CD 45RO, CD4, CD8 and FOXP3(+).

SECONDARY OUTCOMES:
To analyse gastrointestinal toxicity | One week , 2 weeks and 20 days after Metformim beginning
  * To analyse gastrointestinal toxicity grade (examples: nausea, stomach pain, vomiting)
  * Number of Participants with Adverse Events
To analyse the blood tests one day before the biopsy and one day before the surgery | 5 days after blood collection
  -To collect and analyze pre- and post-treatment peripheral blood specimens for serum glucose, glycosylated haemoglobin and insulin levels, as well as circulating IGF-1 and estradiol

CONTACTS AND LOCATIONS:
Overall Officials: Ana Elisa Lohmann, MD, Principal Investigator — Instituto Nacional de Cancer
Locations (1):
- Hospital do Cancer III, Rio de Janeiro, Rio de Janeiro, Brazil